CLINICAL TRIAL: NCT01525927
Title: Phase II Trial of Neoadjuvant Chemotherapy for HPV-Associated Squamous Cell Carcinoma of the Oropharynx Followed by Reduced Dose Radiotherapy/Chemoradiotherapy for Responders or Standard Dose Chemoradiotherapy for Non-Responders
Brief Title: Study of Chemotherapy Prior to Radiotherapy and Chemotherapy in Patients With HPV Associated Cancer of the Oral Cavity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left institution. IRB approval lapsed.
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSLIJ0844
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Oropharyngeal Neoplasms
Keywords: Oropharyngeal Neoplasms; Neoplasms, Oropharyngeal; Oropharynx Neoplasms
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Drug Therapy; Cisplatin; Carboplatin; Etoposide; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy non-responders (Active Comparator): Patients treated with three cycles neoadjuvant chemotherapy who do not exhibit response to chemotherapy are then allocated to recieve standard dose and schedule radiotherapy.
  Interventions: Drug: chemotherapy; Radiation: radiotherapy
- Chemotherapy responders (Experimental): Patients who respond to chemotherapy are treated with reduced dose radiotherapy.
  Interventions: Drug: chemotherapy; Radiation: Reduced dose radiotherapy

INTERVENTIONS:
Drug: chemotherapy — Chemotherapy for three cycles prior to radiotherapy
  Other Names: Cisplatin, Carboplatin, Flourouracil, Etoposide
Radiation: radiotherapy — Standard radiotherapy for non-responders vs reduced dose radiotherapy for responders.
  Other Names: IMRT, Radiation Therapy
  Arms: Chemotherapy non-responders
Radiation: Reduced dose radiotherapy — Patients who achieve a response to chemotherapy then go on to receive reduced dose radiotherapy.
  Other Names: IMRT, Reduced dose radiation therapy
  Arms: Chemotherapy responders

SUMMARY:
This study looks at the use of three cycles of chemotherapy given prior to radiation therapy in patients with cancer of the oral cavity and evidence of prior exposure to Human Papilloma Virus (HPV). Patients with cancer of the oral cavity who have evidence of exposure to HPV have a better prognosis than those who do not have such evidence of exposure to HPV. The main hypothesis of this study is that using three cycles of chemotherapy prior to embarking on radiation therapy will allow the use of reduced doses of radiation therapy and, therefore, less radiation induced side-effects. The primary objective is to determine the activity of this pre-radiation chemotherapy strategy along with reduced dose levels of radiation with or without chemotherapy during the radiation phase. The effectiveness of the strategy will be assessed at three months following the completion of the radiation therapy phase and also at two years following completion of the radiation therapy.

DETAILED DESCRIPTION:
Induction Chemotherapy TPF induction chemotherapy will be administered as published from the TAX 323 phase III trial. Specifically, each cycle will consist of docetaxel at a dose of 75 mg per square meter, administered as a 1-hour infusion on day 1, followed by cisplatin at a dose of 75 mg per square meter, administered as a 1-hour infusion on day 1, and fluorouracil at a dose of 750 mg per square meter per day, administered by continuous infusion on days 1 to 5. Induction chemotherapy will be given every 3 weeks for three cycles, unless there is distant disease progression, unacceptable toxic effects, or withdrawal of consent by the patient. All patients will be required to have a continuous venous access device such as a PICC line or Infusaport type device. This is standard of care for continuous infusion fluorouracil. Response assessment by examination, contrast-enhanced CT imaging and whole body PET-CT will be performed after the third treatment cycle. Radiotherapy or chemoradiotherapy will commence within 3-4 weeks from the conclusion of the induction program.

Selection for Radiation Alone vs. Chemoradiotherapy For CR/PR patients with CR at primary site following induction chemotherapy, locoregional therapy will be risk-adjusted according to baseline tumor stage/characteristics. Local therapy will be 1) radiotherapy as a single modality for Tx (T1-2), T0-1 or exophytic T2, N0-2a disease, or will be 2) concomitant chemoradiotherapy for Tx (T3), endophytic T2, T3, N2b-c disease. Patients with PR at primary site will receive concurrent chemotherapy and reduced dose radiation.

All SD/PD patients will receive concurrent chemotherapy and full dose radiation. Patients catalogued with disease progression on the basis of new distant metastatic disease spread (DM) during induction chemotherapy will be taken off protocol for consideration of palliative therapy.

Concurrent Chemotherapy Concurrent chemotherapy will consist of cisplatin given at 35 mg/m2 weekly for six cycles OR carboplatin given at AUC 1.5 weekly for six cycles. Concurrent chemotherapy will start during the first week of radiation treatment. Selection of either schedule will be left to the discretion of the attending medical oncologist. Concurrent chemotherapy will be held for a platelet count of <100,000 or an absolute neutrophil count of < 1000 per cubic mm.

IMRT doses Primary Target (residual gross disease): 66 Gy called CTV1 (2.2 Gy/fraction in 30 fractions).

Intermediate-Risk Target: 57 Gy called CTV2 (1.9 Gy/fraction in 30 fractions). Prophylactic Target Coverage: 54 Gy called CTV3 (1.8 Gy/fraction in 30 fractions).

IMRT planning Treatment planning CT scans will be required to define target volumes. The treatment planning CT scan should be acquired with the patient in the same position and immobilization device as for treatment. All tissues to be irradiated must be included in the CT scan. MRI or whole body PET/CT scans may be included to assist in definition of target volumes, especially when primary or retropharyngeal nodal disease extends near the base of skull. The immobilization device should include neck and shoulder immobilization. GTV, CTVs, PTVs, and normal tissues must be outlined on all CT slices in which these structures exist.

Primary Target CTV1: All regions of GTV-R in PR patients will receive 66 Gy in 30 fractions, with no attempt to cover remainder of initial GTV. There will be no CTV1 in CR patients.

Intermediate-Risk Target CTV2: This volume encompasses all initial primary and nodal GTV volumes, regions adjacent to GTV (e.g. contralateral base of tongue), as well as complete anatomic coverage of involved cervical neck levels. This will receive 57 Gy in 30 fractions.

Prophylactic Target Coverage CTV3: This volume covers all uninvolved at-risk nodal basins. This will receive 54 Gy in 30 fractions.

Low Neck Conventional Field Treatment: Bilateral low neck/supraclavicular fossae will initially be treated with a beam-split AP field to 40 Gy in 20 fractions with a 3x3 cm larynx block matched at central axis with the inferior edge of IMRT treatment fields. Treatment will then continue to 50 Gy with a midline cord block over 5 daily fractions. Cone-down AP mid neck boosting to 56 Gy will be administered to low neck CTV2, down to the superior edge of the clavicle. Treatment will continue to 64 Gy for low neck CTV1 volumes, respecting brachial plexus dose limitations.

Dose specification The prescription dose is the isodose which encompasses at least 95% of the PTV. No more than 20% of any PTV will receive >110% of its prescribed dose. No more than 1% of any PTV will receive <93% of its prescribed dose. No more than 1% or 1 cc of the tissue outside the PTVs will receive >110% of the dose prescribed to the primary PTV.

Fractionation and treatment duration Treatment will be delivered once daily, 5 fractions per week, over 6 weeks. All targets will be treated simultaneously. Breaks in treatment should be minimized. Break in treatment time of more than 5 days will be considered a major variation and requires documentation underlying the specific reasons for the treatment break (ex. related to study drug and/or chemotherapy and/or RT).

Functional Quality-of-Life Assessments Clinical Assessment of Treatment-Related Symptoms, and Dietary Status: MDASI-HN and MDADI instruments will be self-administered by all study subjects at baseline, treatment completion, and at routine post-radiation surveillance appointments over the subsequent 24 months. At these time points, nutritional status will also be assessed by weight, normalcy of diet score based on the results of the PSS-HN, and feeding tube dependence for any amount of nutritional intake (yes/no). The radiation oncology research nurse will oversee subject completion of these instruments.

MD Anderson Dysphagia Inventory (MDADI): The MDADI measures swallowing-related quality of life (QOL) in patients with swallowing dysfunction. It evaluates the patient's physical, emotional, and functional perceptions of swallowing dysfunction, and has been validated in head and neck cancer patients.

Performance Status Scale for Head and Neck Cancer Patients (PSS-H&N): The PSS-H&N is a clinician rated instrument consisting of three subscales: 1) normalcy of diet, 2) public eating, and 3) understandability of speech. The radiation oncology research nurse or speech-language pathologist will complete the PSS-H&N.

Modified Barium Swallow (MBS) Study: Patients will undergo MBS testing at baseline, 4-6, 12, and 24 months after the completion of ART. Studies will be performed using standard radiographic systems with a videofluoroscope focused on the patient's lips anteriorly, the posterior pharyngeal wall posteriorly, the hard palate superiorly, and the upper esophageal segment inferiorly. The order of bolus presentation will include: two 5-ml Varibar thin liquid boluses, two 10-ml Varibar thin liquid boluses, two 20-ml Varibar thin liquid boluses, two cup sips of Varibar thin liquid, two pureed/Varibar pudding boluses, two solid boluses consisting of ¼ of a shortbread cookie or cracker coated with Varibar pudding, and 2 trials of the most difficult consistency in the A-P plane. The following measures will be used to quantify MBS findings: (1) Penetration-Aspiration Scale (PAS) - The PAS is a clinician rated 8-point, ordinal scale used to describe penetration and aspiration events. Scores are determined by depth of bolus invasion into the airway and the patient's response; a higher score is assumed to be a more severe sign of dysphagia. Intra- and interjudge reliability has been established in head and neck cancer patients. (2) Oropharyngeal swallow efficiency - (OPSE) is a global measure of swallow function defined as the ratio of the percent swallowed into the esophagus divided by oropharyngeal transit time. Thus, a higher OPSE score indicates a safer and more efficient oropharyngeal swallow. The continuous score obtained has been found to correlate with the degree of oropharyngeal dysphagia in head and neck cancer patients. (3) National Institutes of Health Swallowing Safety Scale (NIH-SSS) - The NIH-SSS provides a continuous numeric score to quantify swallowing safety using 7 dysphagia symptoms, residue, penetration, aspiration, response to aspiration, esophageal entry, regurgitation, and multiple swallows. The scale demonstrates high reliability (intra- and interrater intraclass correlation coefficient >.95) and validity in dysphagic patients. We are concurrently evaluating its utility in patients with head and neck cancer. The speech pathologist will complete the PAS, OPSE, and NIH-SSS during analysis of the MBS study.

Salivary Flow Quantification: For unstimulated resting sialometry, each patient will be instructed to first clear the mouth by swallowing. With the head held slightly forward, the patient will be instructed not to swallow during the 5-minute collection, but to allow saliva to collect in the floor of mouth. The patient will expectorate the accumulated saliva into a pre-weighed 100 mL vial after 60 seconds. The patient will repeat this procedure 4 more times for a total collection time of 5 minutes. At the end of the 5 minutes, the collection vial will be promptly sealed and weighed. For each collection, the actual clock time at the start and end of the collection will be recorded as well as the vial weight before and after the collection of the sample. Stimulated sialometry will then be performed. Patients will rest for 5 minutes prior to collection. The exogenous stimulant will be 20 mL of citric acid solution held in the mouth for 1 minute. After the patient expectorates this solution, 5-minute saliva collection will take place as described above. These measurements will be done by the radiation oncology research nurse.

ELIGIBILITY:
Inclusion Criteria:

* Tumor tissue available from primary or nodal metastasis for histological analysis.
* High p16 tumor expression by IHC, or indeterminate p16 expression by IHC and definitively positive detection of high-risk HPV infection by ISH.
* T-stage = T1-3 or post-tonsillectomy Tx (T1-3).
* N-stage = N1-2 or Nx (N1-2).
* Biopsy-confirmed oropharyngeal primary site.
* Histology = squamous cell carcinoma, basaloid-squamous carcinoma, nasopharyngeal-type squamous carcinoma, adenosquamous carcinoma, or papillary squamous carcinoma.
* Age > 17 years old.
* Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count (AGC at least 1500 cells/mm3 and platelet count at least 100,000 cells/mm3); adequate hepatic function with bilirubin less than 1.5x ULN (excluding Gilbert's disease); SGOT, SGPT and alkaline phosphatase must be within the normal range to be eligible for study.
* Creatinine clearance at least 70 ml/min determined by 24 hour collection or nomogram: CrCl male = (140 - age) x (wt in kg)/serum Cr x 72; CrCl female = 0.85 x (CrCl male).
* Patients must have an untransfused hemoglobin of at least 9.0 grams/dL.
* Patients should have no serious acute or chronic co-morbid condition, or acute infection, which in the judgment of the attending physician would affect administration of the induction chemotherapy regimens.
* Patients must sign a study-specific informed consent form.
* All of the above lab criteria must be verified within 28days of registration.

Exclusion Criteria:

* Low p16 expressing tumor by IHC, or indeterminate p16 expression by IHC and negative or weak detection of high-risk HPV infection by ISH.
* TxNx without residual measurable disease, T4, or N3 disease.
* Significant cigarette smoking history, defined as >10 pack-years total lifetime exposure. Pack years is calculated as # packs smoked per day x # years smoking.
* Histology other than squamous cell carcinoma.
* Proven distant metastases (below the clavicle) by clinical or radiographic measures.
* Karnofsky performance status < 80 or ECOG >1.
* Prior chemotherapy, within the previous 3 years.
* Prior radiotherapy to the head and neck.
* Initial surgical resection rendering the patient clinically and radiologically disease free.
* Simultaneous primary invasive cancers, excluding superficial non-melanoma skin cancers.
* Patients with a history of another malignancy (excluding non melanoma skin cancers, and cancers treated > 3 years prior for which patient remains continuously disease free).
* Men and women of childbearing potential (WOCBP) unwilling to consent to using effective contraception while on treatment and for at least 3 months thereafter. Note: WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study and for 3 months after the study in such a manner that the risk of pregnancy is minimized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhoomi Mehrotra, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

REFERENCES:
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Chaturvedi AK, Engels EA, Anderson WF, Gillison ML. Incidence trends for human papillomavirus-related and -unrelated oral squamous cell carcinomas in the United States. J Clin Oncol. 2008 Feb 1;26(4):612-9. doi: 10.1200/JCO.2007.14.1713. PMID 18235120
- [Background] Gillison ML, Koch WM, Capone RB, Spafford M, Westra WH, Wu L, Zahurak ML, Daniel RW, Viglione M, Symer DE, Shah KV, Sidransky D. Evidence for a causal association between human papillomavirus and a subset of head and neck cancers. J Natl Cancer Inst. 2000 May 3;92(9):709-20. doi: 10.1093/jnci/92.9.709. PMID 10793107
- [Background] Herrero R, Castellsague X, Pawlita M, Lissowska J, Kee F, Balaram P, Rajkumar T, Sridhar H, Rose B, Pintos J, Fernandez L, Idris A, Sanchez MJ, Nieto A, Talamini R, Tavani A, Bosch FX, Reidel U, Snijders PJ, Meijer CJ, Viscidi R, Munoz N, Franceschi S; IARC Multicenter Oral Cancer Study Group. Human papillomavirus and oral cancer: the International Agency for Research on Cancer multicenter study. J Natl Cancer Inst. 2003 Dec 3;95(23):1772-83. doi: 10.1093/jnci/djg107. PMID 14652239
- [Background] Hashibe M, Brennan P, Benhamou S, Castellsague X, Chen C, Curado MP, Dal Maso L, Daudt AW, Fabianova E, Fernandez L, Wunsch-Filho V, Franceschi S, Hayes RB, Herrero R, Koifman S, La Vecchia C, Lazarus P, Levi F, Mates D, Matos E, Menezes A, Muscat J, Eluf-Neto J, Olshan AF, Rudnai P, Schwartz SM, Smith E, Sturgis EM, Szeszenia-Dabrowska N, Talamini R, Wei Q, Winn DM, Zaridze D, Zatonski W, Zhang ZF, Berthiller J, Boffetta P. Alcohol drinking in never users of tobacco, cigarette smoking in never drinkers, and the risk of head and neck cancer: pooled analysis in the International Head and Neck Cancer Epidemiology Consortium. J Natl Cancer Inst. 2007 May 16;99(10):777-89. doi: 10.1093/jnci/djk179. PMID 17505073
- [Background] Fakhry C, Westra WH, Li S, Cmelak A, Ridge JA, Pinto H, Forastiere A, Gillison ML. Improved survival of patients with human papillomavirus-positive head and neck squamous cell carcinoma in a prospective clinical trial. J Natl Cancer Inst. 2008 Feb 20;100(4):261-9. doi: 10.1093/jnci/djn011. Epub 2008 Feb 12. PMID 18270337
- [Background] Carvalho AL, Nishimoto IN, Califano JA, Kowalski LP. Trends in incidence and prognosis for head and neck cancer in the United States: a site-specific analysis of the SEER database. Int J Cancer. 2005 May 1;114(5):806-16. doi: 10.1002/ijc.20740. PMID 15609302
- [Background] Hafkamp HC, Manni JJ, Haesevoets A, Voogd AC, Schepers M, Bot FJ, Hopman AH, Ramaekers FC, Speel EJ. Marked differences in survival rate between smokers and nonsmokers with HPV 16-associated tonsillar carcinomas. Int J Cancer. 2008 Jun 15;122(12):2656-64. doi: 10.1002/ijc.23458. PMID 18360824
- [Background] Shiboski CH, Schmidt BL, Jordan RC. Tongue and tonsil carcinoma: increasing trends in the U.S. population ages 20-44 years. Cancer. 2005 May 1;103(9):1843-9. doi: 10.1002/cncr.20998. PMID 15772957
- [Background] Sturgis EM, Cinciripini PM. Trends in head and neck cancer incidence in relation to smoking prevalence: an emerging epidemic of human papillomavirus-associated cancers? Cancer. 2007 Oct 1;110(7):1429-35. doi: 10.1002/cncr.22963. PMID 17724670
- [Background] Garden AS, Asper JA, Morrison WH, Schechter NR, Glisson BS, Kies MS, Myers JN, Ang KK. Is concurrent chemoradiation the treatment of choice for all patients with Stage III or IV head and neck carcinoma? Cancer. 2004 Mar 15;100(6):1171-8. doi: 10.1002/cncr.20069. PMID 15022283
- [Background] Mork J, Lie AK, Glattre E, Hallmans G, Jellum E, Koskela P, Moller B, Pukkala E, Schiller JT, Youngman L, Lehtinen M, Dillner J. Human papillomavirus infection as a risk factor for squamous-cell carcinoma of the head and neck. N Engl J Med. 2001 Apr 12;344(15):1125-31. doi: 10.1056/NEJM200104123441503. PMID 11297703
- [Background] D'Souza G, Kreimer AR, Viscidi R, Pawlita M, Fakhry C, Koch WM, Westra WH, Gillison ML. Case-control study of human papillomavirus and oropharyngeal cancer. N Engl J Med. 2007 May 10;356(19):1944-56. doi: 10.1056/NEJMoa065497. PMID 17494927
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Dahlstrom KR, Adler-Storthz K, Etzel CJ, Liu Z, Dillon L, El-Naggar AK, Spitz MR, Schiller JT, Wei Q, Sturgis EM. Human papillomavirus type 16 infection and squamous cell carcinoma of the head and neck in never-smokers: a matched pair analysis. Clin Cancer Res. 2003 Jul;9(7):2620-6. PMID 12855639
- [Background] Laccourreye O, Brasnu D, Bassot V, Menard M, Khayat D, Laccourreye H. Cisplatin-fluorouracil exclusive chemotherapy for T1-T3N0 glottic squamous cell carcinoma complete clinical responders: five-year results. J Clin Oncol. 1996 Aug;14(8):2331-6. doi: 10.1200/JCO.1996.14.8.2331. PMID 8708725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants enrolled, no data collected, no documentation of study intervention.
Period: Overall Study
Arm/Group | Chemotherapy Responders
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: data was not collected for Baseline Characteristics due to premature termination of this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Non-responders | Chemotherapy Responders | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Response (CR+PR) Status at 3 Months Post-therapy
Description: The 3-month response rate will be estimated using standard methods for estimating proportions and their 95% one-sided confidence intervals (CIs). Comparison to the historical control data will be carried out using a chi-square test for comparing proportions (or a Fisher exact test if an expected cell frequency in the 2x2 table is less than 5).
  Zero (0) participants analyzed
Time Frame: 3 months following completion of radiation phase
Population: No study intervention or data collected.
Arm/Group | Chemotherapy Responders
Number analyzed (Participants) | 0

2. Secondary Outcome: To Define Objective Tumor Response Rates to Induction Chemotherapy and to Subsequent Radiation-based Treatment.
Description: To define objective tumor response rates to induction chemotherapy and to subsequent radiation-based treatment, per RESIST version 1.1 criteria.
Time Frame: Three months following completion of radiation therapy phase.
Groups:
- No Study Intervention or Data Collected- Zero (0) Participants: No study intervention or data collected- Zero (0) participants analyzed
Arm/Group | No Study Intervention or Data Collected- Zero (0) Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival at 2 Years
Description: assess Progression-free survival at 2 years.
Time Frame: At two years following completion of radiation phase
Population: No study intervention or data collected- Zero (0) participants analyzed
Arm/Group | No Study Intervention or Data Collected- Zero (0) Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Assess Overall Survival at 2 Years.
Description: To assess overall survival at 2 years.
Time Frame: At two years following completion of radiation phase
Population: No study intervention or data collected- Zero (0) participants analyzed
Arm/Group | No Study Intervention or Data Collected- Zero (0) Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Assess Locoregional Disease Control at 2 Years
Description: To assess locoregional disease control at 2 years
Time Frame: At two years following completion of radiation phase
Population: No study intervention or data collected- Zero (0) participants analyzed
Arm/Group | No Study Intervention or Data Collected- Zero (0) Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Assess Distant Disease Control at 2 Years.
Description: 3.5 To assess distant disease control at 2 years.
Time Frame: At two years following completion of radiation phase
Population: No study intervention or data collected- Zero (0) participants analyzed
Arm/Group | No Study Intervention or Data Collected- Zero (0) Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Assessment of Quality of Life Outcomes
Description: Serial evaluation of functional quality-of-life, including M. D. Anderson Dysphagia Inventory (MDADI) and Oropharyngeal swallowing efficiency (OPSE) measures of swallowing function, as well as formal sialometric measurement of parotid function.
Time Frame: Baseline, during therapy and up to two years following completion of radiation phase
Population: No study intervention or data collected- Zero (0) participants analyzed
Arm/Group | No Study Intervention or Data Collected- Zero (0) Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Identify Additional Toxicity of Treatment
Description: To identify additional toxicity of treatment
Time Frame: During therapy and up to 5 years following completion of treatment
Population: No study intervention or data collected- Zero (0) participants analyzed
Arm/Group | No Study Intervention or Data Collected- Zero (0) Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed due to premature termination of this study.
Groups:
- Chemotherapy Non-responders: Patients treated with three cycles neoadjuvant chemotherapy who do not exhibit response to chemotherapy are then allocated to recieve standard dose and schedule radiotherapy.
  chemotherapy: Chemotherapy for three cycles prior to radiotherapy
  radiotherapy: Standard radiotherapy for non-responders vs reduced dose radiotherapy for responders.
  Zero (0) participants analyzed
- Chemotherapy Responders: Patients who respond to chemotherapy are treated with reduced dose radiotherapy.
  chemotherapy: Chemotherapy for three cycles prior to radiotherapy
  Reduced dose radiotherapy: Patients who achieve a response to chemotherapy then go on to receive reduced dose radiotherapy.
  Zero (0) participants analyzed
Arm/Group | Chemotherapy Non-responders | Chemotherapy Responders
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated , PI left the institution, no data analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes